CLINICAL TRIAL: NCT04057066
Title: Internet-based Physical Activity Promotion and Exercise Prescription for People With Multiple Sclerosis. A Feasibility Study.
Brief Title: Internet-based Physical Activity Promotion and Exercise Prescription for People With Multiple Sclerosis (Feasibility Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: Neurological Rehabilitation Center Quellenhof (Unknown); ZTM Bad Kissingen (Other); Medi train - Zentrum für Gesundheitssport, Sport- und Physiotherapie (Unknown); proMX GmbH Nürnberg (Unknown); motionNET systems Limited (Unknown); Aktion Multiple Sklerose Erkrankter, Landesverband der DMSG in Baden-Württemberg (AMSEL) e.V. (Unknown); Klinikum Würzburg Mitte GmbH (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Head of the Department of Sport Science and Sport, University of Erlangen-Nürnberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ms bewegt 1.2
Record Dates: First submitted 2019-08-08; First posted 2019-08-14 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; e-health; physical activity promotion; exercise; feasibility; online; internet based
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants receive physical activity counseling as well as an individualized exercise plan.
  Interventions: Behavioral: Physical activity counseling; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Physical activity counseling — Physical activity counseling consists of two phone or video calls with a therapists, two group video calls with a therapist and a complementary e-learning course.
Behavioral: Exercise — Participants will agree with their therapist on an exercise plan (endurance and resistance training) that will be made available through the studies mobile app. Frequency and duration of endurance and strength training shall be prescribed in accordance with exercise guidelines for pwMS. However, they can be adjusted according to participants prior physical activity level and their available time slots for exercise during the week.

SUMMARY:
This study evaluates the feasibility of a 12-week internet-based exercise and physical activity counseling intervention for people with Multiple Sclerosis (MS).

DETAILED DESCRIPTION:
Due to high inactivity rates in persons with Multiple Sclerosis (pwMS) physical activity promotion for this target group is needed. The internet is an attractive and feasible medium for physical activity promotion, however interventions have to be adapted to the special needs of pwMS. This study aims to evaluate the feasibility of a 12-week internet-based exercise and physical activity counseling intervention.

26 pwMS will be enrolled in the study. All of them receive the intervention. Focus groups and interviews will be conducted with participating pwMS to determine acceptability of the intervention and to explore participants experiences. Compliance with the intervention will be monitored. Additionally, changes in objective physical activity, subjective physical activity, fatigue, walking ability and level of depression will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed Multiple Sclerosis (McDonald criteria)
* expanded Disability Status Scale between 0 - 6.5
* neurologically stable (no exacerbation within 30 days prior to enrollment)
* internet access (WiFi)
* basic knowledge on handling personal computer and the internet
* owning a smartphone with the operating system Android or IOS and with access to Google Play Store or Apple App score
* ability to read, write and comprehend as well as communicate electronically
* not regularly physically active (more than 30 minutes twice a week with a moderate intensity (includes aerobic training, resistance training and other sports e.g. Tennis; excludes physiotherapy, physical activity during work or household, grocery shopping, gardening, walking the dog etc.)

Exclusion Criteria:

* clinically relevant cardiovascular diseases
* cortisone therapy in the last 30 days
* cognitive impairment
* severe impairment of hand function (ataxia or paresis impeding the use of a smartphone app or smartwatch)
* severe internal, orthopaedic and metabolic diseases that restrict mobility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Acceptability of the Intervention and participants' experiences (focus groups) | 1 week after the end of the intervention
  Focus groups (1,5 hrs) with participants to determine extent to which they perceived intervention as appropriate.
Compliance with intervention protocol (completed training sessions and e-learning modules) | over the 12 weeks of intervention
  Completed training sessions and e-learning modules will be documented for each participant with the interventions mobile app and e-learning course.
Acceptability of the Intervention and participants' experiences (interviews) | 1 week after the end of the intervention
  With those participants that cannot take part in the focus groups, semistructured interviews (30 min) will be conducted to determine extent to which participants' perceived intervention as appropriate. Interview questions are based on focus group questions. The wording is slightly adapted to fit the interview situation.

SECONDARY OUTCOMES:
Changes in objectively measures physical activity | 1 week before start of the intervention (T0), 1 week after the end of the intervention (T1)
  The physical activity level of participants is measured over a 7 day period with the accelerometer Actigraph GT3X+. The Actigraph GT3X+ measures acceleration on three axes. Steps per day, physical activity per day (activity counts) and time in moderate and vigorous physical activity per day will be calculated.
Changes in subjectively measured physical activity: European Health Interview Survey-Physical Activity Questionnaire (EHIS-PAQ) | 1 week before start of the intervention (T0), 1 week after end of the intervention (T1)
  8-item questionnaire to assess time spent for work related physical activity, physical activity for transportation (walking, biking), muscle strengthening exercises and sports, fitness or recreational physical activity during a typical week.
Würzburger Fatigue Inventory for MS (WEIMuS) | 1 week before start of the intervention (T0), 1 week after the end of the intervention (T1)
  This questionnaire contains 17 items that form a physical and cognitive subscale. The total score ranges from zero to a maximum of 68 points (maximum fatigue). The cut-off value for the presence of fatigue is above 32.
Allgemeine Depressionsskala (ADS-L) | 1 week before start of the intervention (T0), 1 week after the end of the intervention (T1)
  German version of the Center for Epidemiologic Studies Depression Scale, 20 item questionnaire. Each item is rated on a 4-point Likert scale. Answers are scored from 0 to 3. The scores for all items are added up to receive the total score. The total score ranges from 0 to 60 with higher scores representing higher levels of depression.
Multiple Sclerosis Walking Scale-12 | 1 week before start of the intervention (T0), 1 week after the end of the intervention (T1)
  12-item questionnaire measuring self reported walking ability. Each item is answered on a 5-point Likert scale. Answers are scored from 1 to 5. The scores for all items are added up to receive a total score. The total score ranges from 12 to 60 with higher scores representing higher levels of depression. As a last step the total score is transformed into the walk12-score ranging from 0 to 100 ((total score -12)/48 x 100 = walk12-score).

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Pfeifer, Prof. Dr., Principal Investigator — Friedrich-Alexander-Universität Erlangen-Nürnberg, Department of Sport Science and Sport; Peter Flachenecker, Prof. Dr. med., Principal Investigator — Neurological Rehabilitation Center Quellenhof; Mathias Mäurer, Prof. Dr. med., Principal Investigator — Klinikum Würzburg Mitte gGmbH
Locations (3):
- Germany (3):
  - Neurological Rehabilitation Center Quellenhof, Bad Wildbad, Baden-Wurttemberg
  - Klinikum Würzburg Mitte gGmbH, Würzburg, Bavaria
  - Friedrich-Alexander-Universität Erlangen-Nürnberg (FAU), Erlangen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Official description of the project on the website of the University of Erlangen-Nürnberg. — https://www.sport.fau.de/ms-bewegt/